CLINICAL TRIAL: NCT02037607
Title: Incidence of Venous Thromboembolism in Children Undergoing Elective Neurosurgical Procedures
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Daniel Fulkerson, Neurosurgeon, Indiana University
Other Study IDs: 1208009386
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Children; Pediatric; Anti-coagulant; Neurosurgical procedures; Blood Clot
MeSH Terms: conditions — Venous Thrombosis; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine how frequently children undergoing elective neurosurgical procedures develop blood clots in the deep veins of the legs while hospitalized. The information gained from this study will help us determine when children children need to receive therapy to help prevent this type of blood clot from forming.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 1 month-12 years undergoing elective neurosurgical procedures.

Exclusion Criteria:

* Patients undergoing outpatient neurosurgical procedures
* Patients with known DVT
* Patients with known hypercoagulable state
* Patients at high risk for DVT (discretion of surgeon in consultation with the hematology service)

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100 children between the ages of 1 month-12 years having an elective neurosurgical procedure at James Whitcomb Riley Hospital for Children.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Fulkerson, M.D., Principal Investigator — Indiana University
Locations (1):
- James Whitcomb Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Scherer AG, White IK, Shaikh KA, Smith JL, Ackerman LL, Fulkerson DH. Risk of deep venous thrombosis in elective neurosurgical procedures: a prospective, Doppler ultrasound-based study in children 12 years of age or younger. J Neurosurg Pediatr. 2017 Jul;20(1):71-76. doi: 10.3171/2017.3.PEDS16588. Epub 2017 May 5. PMID 28474980

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound Group (All): All subjects in the study are in the same group. Study procedure is ultrasound
Period: Overall Study
Arm/Group | Ultrasound Group (All)
Started | 100
Completed | 91
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: 91 subjects received study procedures and were analyzed. 9 additional subjects were consented but withdrawn prior to completion of study procedures.
Groups:
- Ultrasound Group (All): All subjects in the study are in the same group. Study procedure is ultrasound within 48 hours prior to surgery and a repeat within 72 hours after surgery.
Arm/Group | Ultrasound Group (All)
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 91
Received baseline ultrasound [Count of Participants; unit: Participants] | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-operative Ultrasound Without Evidence of Thromboembolism
Description: The number of participants with post-operative ultrasound without evidence of thromboembolism
Time Frame: within 72 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Group (All)
Number analyzed (Participants) | 91
Participants | 91

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected as this was a minimal risk study
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Ultrasound Group (All)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes